CLINICAL TRIAL: NCT00311454
Title: An Open Single Centre Evaluation of the Reactivity of the T.R.U.E. Test Quaternium-15 Patch and a Real Use Exposure in Subjects Known to Be Allergic to Quaternium-15
Brief Title: Quaternium-15, Use Test
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mekos Laboratories AS (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Mekos 05 UseQ 001
Record Dates: First submitted 2006-04-04; First posted 2006-04-06 (Estimated); Last update posted 2006-04-06 (Estimated); Status verified 2006-04

CONDITIONS: Allergic Contact Dermatitis Towards Quaternium-15

INTERVENTIONS:
Drug: T.R.U.E.Test

SUMMARY:
The study is required by the FDA as part of a post-marketing commitment. The purpose of the study is to compare the reactivity of the TRUE Test quaternium-15 patch and a real use exposure.The subjects will wear the patch test for 48 hours and reading will be performed day 3 or 4. The use test will be applied from day 3 or 4 and untill reaction appears. Reactions from respectively TRUE Test and use test will be compared using the McNemar Change Test.

ELIGIBILITY:
Inclusion Criteria:

* Sensitivity to quaternium-15
* Age more than 18 years

Exclusion Criteria:

* Topical or systemic treatment with corticosteroids or immunosuppresives.
* Treatment with UV-light
* Widespread active dermatitis or dermatitis on test area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2006-04

CONTACTS AND LOCATIONS:
Locations (1):
- Amtssygehuset i Gentofte, Gentofte Municipality, Gentofte, Denmark